CLINICAL TRIAL: NCT05272293
Title: Immunotherapy With ex Vivo Expanded Haploidentical Natural Killer Cells for Children/Young Adults With High-risk, Refractory or Relapsed AML
Brief Title: Immunotherapy With ex Vivo Expanded Haploidentical Natural Killer Cells for Children/Young Adults With AML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Belarusian Research Center for Pediatric Oncology, Hematology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: haploNK_ HR/R/R_AML
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Natural killer cells, immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- expanded haploidentical NK cell immunotherapy (Experimental): After a cycle of chemotherapy a patient receive three intravenous infusions of expanded haploidentical NK cells.
  Interventions: Biological: NK cell infusions

INTERVENTIONS:
Biological: NK cell infusions — Three doses of expanded haploidentical NK cells (30-100 x 10^6 cells /kg).

SUMMARY:
The purpose of this study is to estimate the efficacy of immunotherapy with ex vivo expanded haploidentical NK cells for children/young adults with primary high risk or refractory AML and relapsed AML.

DETAILED DESCRIPTION:
Immunotherapy with NK cells may improve the treatment results in AML. For better efficiency high cell doses or several infusions of NK cells are required. For this purpose, donor NK cells are expanded in the presence of feeder K562-mbIL21-41BBL cell line.

For patients with high-risk primary AML a cycle of immunotherapy includes chemotherapy (HD-ARA-C+IDA) followed by three doses of NK cells infusion.

For patients with refractory/relapsed AML a cycle of immunotherapy includes chemotherapy (FLAG - fludarabine, cytarabine, G-CSF) followed by three doses of NK cells infusion.

A 2nd cycle of therapy may be administered if a recipient continues to meet the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* primary high risk AML
* primary refractory AML
* relapsed AML
* Karnofsky or Lansky performance scale greater or equal to 70
* written informed consent

Donors:

* haploidentical family donor
* donor suitable for cell donation and apheresis according to standard criteria
* written informed consent

Exclusion Criteria:

Patients:

* uncontrolled infection
* severe hepatic dysfunction: SGOT or SCPT >=5x upper limit of normal for age
* positive serology for human immunodeficiency virus (HIV)

Donors:

* pregnancy
* positive serology for HIV, hepatitis B or C

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) (PR+ MLFS+CRi +CR) | 30 days after every a course of NK immunotherapy
  The proportion of patients with complete remission (CR), CR with incomplete hematologic recovery (CRi), morphologic leukemia-free state (MLFS), and partial remission (PR) as measured by response criteria definitions for acute myeloid leukemia.
Leukemia-free survival (LFS) | 1 year
  Time from achievement of CR/CRi/MLFS to the time of relapse, death in remission, or last follow-up.
Overall survival (OS) | 1 year
  The proportion of patients with overall survival

SECONDARY OUTCOMES:
Duration of persistence of infused NK cells | 21 days after the first infusion
  Days of persistence of donor NK cells
Number of T, B, NK, activated T and NK cells after immunotherapy | 30 days after the first infusion
  Analysis of T, B, NK, activated T and NK cells numbers (cells/microL) after NK infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Aleinikova, MD, Prof, Principal Investigator — Belarussian Research Center for Pediatric Oncology, Hematology and Immunology
Locations (1):
- Belarussian Research Center for Pediatric Oncology, Hematology and Immunology, Minsk, Minsk Oblast, Belarus